CLINICAL TRIAL: NCT02034084
Title: A Comparison of Left and Right Radial Approach for Percutaneous Coronary Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Buxing Chen, Director of department of cardiology, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COLAR
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2014-01

CONDITIONS: Transradial Approach,; Coronary Angiography,; Percutaneous Coronary
Keywords: Transradial approach,; Coronary angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Right radial approach (Experimental): Coronary diagnostic procedures performed through right radial approach
  Interventions: Procedure: Right radial approach
- Left radial approach (Experimental): Coronary diagnostic procedures performed through left radial approach
  Interventions: Procedure: left radial approach

INTERVENTIONS:
Procedure: left radial approach — Coronary diagnostic procedures performed through left radial approach
  Arms: Left radial approach
Procedure: Right radial approach — coronary diagnostic procedures performed through right radial approach
  Arms: Right radial approach

SUMMARY:
Previous studies have shown that the transradial cardiac catheterization has decreased not only bleeding complications related to the access site and procedural discomfort but also morbidity and hospitalization as compared to transfemoral approach. At present, the right radial approach (RRA) is the first choice routinely for coronary angiography and interventions in daily clinical practice despite more marked subclavian artery tortuosity than left radial approach (LRA). Although LRA has been thought to be more direct access to the ascending aorta similar to transfemoral approach and may reduce fluoroscopy time and cerebrovascular complications compared with RRA, the application of LRA for coronary intervention is still low. Moreover, several studies have also obtained conflicting results showing no difference in procedural success rate compared LRA and RRA using Judkins catheters. To date, it remains unclear whether LRA is superior to RRA in term of safety and feasibility for coronary angiography and interventions in real world practice and few data of randomized control trial are available.

The aim of this study was to randomly investigate and compare the safety and feasibility of LRA compared with RRA for coronary diagnostic angiography in Chinese subjects.

The investigators will enroll consecutively for 2 years all patients undergoing coronary diagnostic procedures through trans radial approach.

The primary outcome was total procedural duration. Secondary outcomes included fluoroscopy time, dose of radiation including cumulative air kerma and dose area product, contrast volume and the incidence of vascular complications.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients who undergo to diagnostic coronary procedures

Exclusion Criteria:

* Acute ST-elevation myocardial infarction
* Previous coronary artery bypass graft surgery
* Hemodynamic instability

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Actual)
Dates: Start 2011-03; Primary Completion 2013-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Total procedural duration | 1 day

SECONDARY OUTCOMES:
Fluoroscopy time | 7 days
Dose of radiation | 7 days
  Dose of radiation include cumulative air kerma (CAK) and CAK dose area product (CAK DAP)
Contrast volume | 7 days

OTHER OUTCOMES:
Vascular complications | 7 days
  Vascular complications include stroke, pseudoaneurysm, arteriovenous fistula, lose of radial artery pulse, puncture site bleeding and forearm hematoma.

CONTACTS AND LOCATIONS:
Overall Officials: Buxing Chen, Dr, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China